CLINICAL TRIAL: NCT05815056
Title: Comparaison Between Virtual Reality Hypnosis and Drug Induced Sedation in Veinous Access Device Implantation
Brief Title: Comparaison Between Digital and Drug Induced Sedation in Veinous Access Device Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Regional de Huy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022 PAC RV vs sed med
Record Dates: First submitted 2023-02-06; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Oncology
Keywords: central veinous catheter; virtual reality induced hypnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 1 arm with anaesthetic drugs vs hypnosis induced by virtual reality
Masking Description: the participation in one of the 2 arms is determined randomly just before the implantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug intervention (Active Comparator): drug induced sedation
  Interventions: Drug: drug intervention
- digital sedation (Experimental): hypnosis induced by a virtual reality device
  Interventions: Device: Sedakit (R) using hypnosis induced by the virtual reality device

INTERVENTIONS:
Device: Sedakit (R) using hypnosis induced by the virtual reality device — we use the virtual reality device and no medication during the surgery
  Other Names: Oncomfort
  Arms: digital sedation
Drug: drug intervention — using sufentanyl 5mg intravenously during the surgery
  Other Names: medical sedation
  Arms: drug intervention

SUMMARY:
The goal of this clinical trial is to compare in patients who need an implantation of a veinous access device the sedation with anesthesiologic drugs and with hypnosis using virtual reality material. The main question it aims to answer is:

• is hypnosis using virtual reality as safe and powerfull than usual anesthesiologic drugs.

Participants will complete a preoperative and postoperative questionnaire. They will be contacted by phone pre and postoperatively.

If there is a comparison group: Researchers will compare drug induced sedation and hypnosis induced by virtual reality to see if they are similar in efficacy and sides effects.

DETAILED DESCRIPTION:
This study has two arms. All patients has the same preparation to surgery. They had lorazepam 2.5 mg 30 minutes before the surgery. In operative theater, they are randomly chosen between anesthetic protocol (sufentanyl 5mg intravenous) or digital sedation (Sedakit(R) ) with hypnosis induced by virtual reality.

Patients complete an anxiety test (hamilton scale) 2 days before the surgery and 2 days after the surgery. They are called by an external psychiatrist 1 day before the surgery and 3 days after to evaluate the anxiety link to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* need for a venous device implantation

Exclusion Criteria:

* need for a general anaesthesia
* unability to give oral consent
* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
successful implantation of a veinous access device | immediately after surgery
  we evaluate if the veinous access was implanted successfully with digital or drug sedation

SECONDARY OUTCOMES:
patient comfort | during the surgery
  we evaluate if the patient needed additional pain killers during the procedure
implantation lenght | during the surgery
  we evaluate the length of the implantation in minutes with the drug or digital sedation
feeling lenght | immediately after the surgery
  we evaluate the length of the implantation felt by the patient using drug or digital sedation
post operative anxiety using the hamilton anxiety scale | 2 days after the surgery
  we do a post operative test to evaluate the level of anxiety after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: JeanFrancois Maillart, MD, Principal Investigator — CHR de Huy
Locations (1):
- CHR de Huy, Huy, Belgium

IPD SHARING:
Plan to Share IPD: Yes
an article will be published with the results. the results will probably be exposed in a future congress.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: the data will be available after the official publication for one year
Access Criteria: official asking and scientific interest in this study.